CLINICAL TRIAL: NCT03091790
Title: Mesh Type in Ventral Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Julie Holihan, Staff Physician, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSC-MS-16-0936
Record Dates: First submitted 2017-03-21; First posted 2017-03-27 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Ventral Hernia
Keywords: ventral hernia; mesh
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Synthetic Mesh (Active Comparator): Synthetic mesh (mid-density polypropylene (generic) Bard soft mesh) will be used in open ventral hernia repair
  Interventions: Device: Synthetic Mesh
- Biologic Mesh (Active Comparator): Biologic mesh (non cross linked porcine acellular dermal matrix: Strattice) will be used in open ventral hernia repair
  Interventions: Device: Biologic Mesh

INTERVENTIONS:
Device: Synthetic Mesh — Synthetic mesh used during open ventral hernia repair
  Arms: Synthetic Mesh
Device: Biologic Mesh — Biologic mesh used during open ventral hernia repair
  Arms: Biologic Mesh

SUMMARY:
Ventral hernias are common following abdominal surgery. Currently, there is no equipoise on when synthetic and biologic meshes should be used. Among open ventral hernia repairs, half are repaired using biologic mesh while half are repaired using synthetic mesh. The investigators hypothesize that biologic mesh as opposed to synthetic mesh repair of open ventral hernia repair is associated with decreased risk of major complications one year after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled for open ventral hernia repair at LBJ General Hospital

Exclusion Criteria:

* Active infection
* Patient unlikely to survive with the next 2 years based upon surgeon judgment (i.e. metastatic cancer, end-stage cirrhosis)
* Patient surgeon would not normally place a prosthetic (e.g. planned second surgery such as ostomy takedown)
* Patient unlikely to follow-up (i.e. no phone)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2020-07-26 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Complication free at 1 year post-operative | 1 year after surgery
  Complication defined as hernia recurrence, chronic wound complications including mesh infection, and reoperation

SECONDARY OUTCOMES:
Complication free at 3 years post-operative | 3 years after surgery
  Complication defined as hernia recurrence, chronic wound complications including mesh infection, and reoperation
Dindo-clavien complications | Pre-operative, 1 month after surgery, 1 year and 3 years after surgery
  Grade I to V
Patient centered outcomes | Pre-operative, 1 month after surgery, 1 year and 3 years after surgery
  includes patient satisfaction, cosmetic satisfaction, modified assessment scale
Cost | 1 year and 3 years after surgery
  charges for all patient visits, admissions, and procedures

CONTACTS AND LOCATIONS:
Overall Officials: Julie L Holihan, M.D., Principal Investigator — UT Health
Locations (1):
- UT Health at Lyndon B. Johnson General Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided